CLINICAL TRIAL: NCT01193842
Title: A Sequential Phase I/Randomized Phase II Trial of Vorinostat and Risk-Adapted Chemotherapy With Rituximab in HIV-Related B-Cell Non-Hodgkin's Lymphoma
Brief Title: Vorinostat and Combination Chemotherapy With Rituximab in Treating Patients With HIV-Related Diffuse Large B-Cell Non-Hodgkin Lymphoma or Other Aggressive B-Cell Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02508; NCI-2011-02508 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000683379; AMC #75; AMC-075 (Other: AIDS Malignancy Consortium); AMC-075 (Other: CTEP); UM1CA121947 (NIH)
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-10

CONDITIONS: AIDS-Related Plasmablastic Lymphoma; AIDS-Related Primary Effusion Lymphoma; Ann Arbor Stage I Diffuse Large B-Cell Lymphoma; Ann Arbor Stage I Grade 3 Follicular Lymphoma; Ann Arbor Stage II Diffuse Large B-Cell Lymphoma; Ann Arbor Stage II Grade 3 Contiguous Follicular Lymphoma; Ann Arbor Stage II Grade 3 Non-Contiguous Follicular Lymphoma; Ann Arbor Stage III Diffuse Large B-Cell Lymphoma; Ann Arbor Stage III Grade 3 Follicular Lymphoma; Ann Arbor Stage IV Diffuse Large B-Cell Lymphoma; Ann Arbor Stage IV Grade 3 Follicular Lymphoma; HIV Infection; Plasmablastic Lymphoma; Primary Effusion Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Grade 3 Follicular Lymphoma
MeSH Terms: conditions — HIV Infections; Plasmablastic Lymphoma; Lymphoma, Primary Effusion; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — Cyclophosphamide; Doxorubicin; Etoposide; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (VR-DA-EPOCH) (Experimental): Patients receive vorinostat PO QD on days 1-5; rituximab IV on day 1; etoposide IV over 24 hours, doxorubicin hydrochloride IV over 24 hours, and vincristine sulfate IV over 24 hours on days 1-4; prednisone PO daily on days 1-5; and cyclophosphamide IV over 1 hour on day 5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate; Drug: Vorinostat
- ARM B (DA-R-EPOCH) (Experimental): Patients receive rituximab, etoposide, doxorubicin hydrochloride, vincristine sulfate, prednisone, and cyclophosphamide as in Arm A. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza
  Arms: Arm A (VR-DA-EPOCH)

SUMMARY:
This partially randomized phase I/II trial studies the side effects and the best dose of vorinostat when given together with combination chemotherapy and rituximab to see how well it works compared to combination chemotherapy alone in treating patients with human immunodeficiency virus-related diffuse large B-cell non-Hodgkin lymphoma or other aggressive B-cell lymphomas. Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as rituximab, may interfere with the ability of cancer cells to grow and spread. Giving vorinostat together with combination chemotherapy and rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the recommended phase II dose (RPTD) of vorinostat that may be used in combination with dose-adjusted etoposide, prednisone, vincristine sulfate, cyclophosphamide, doxorubicin hydrochloride and rituximab (R-DA-EPOCH) (in high-risk disease) in participants with human immunodeficiency virus (HIV)-associated aggressive cluster of differentiation (CD)20 positive non-Hodgkin lymphoma (NHL). (Phase I) II. Determine the overall toxicity rates of R-DA-EPOCH (in high-risk disease) with and without vorinostat. (Phase II) III. Determine the efficacy of the combinations of R-DA-EPOCH (in high-risk disease) with and without vorinostat in HIV-associated aggressive CD20 positive NHL using complete response (CR) rates as study endpoints. (Phase II)

SECONDARY OBJECTIVES:

I. Determine 1-year event-free survival (EFS) and 1 year overall survival (OS). II. Assess the effect of vorinostat and chemotherapy on latent HIV in memory T cells.

III. Assess the effect of vorinostat and/or chemotherapy on HIV, Epstein-Barr virus (EBV), and human herpes virus 8 (HHV-8) viral loads on banked specimens.

IV. Assess the effect of vorinostat and/or chemotherapy on T-cell subsets (CD4 and CD8) and plasma immunoglobulin levels.

V. Assess the effect of concurrent vorinostat and rituximab on plasma steady-state concentrations of etoposide, doxorubicin (doxorubicin hydrochloride), and vincristine (vincristine sulfate) (on Phase I only).

VI. Perform wide human gene expression profiling and methylation studies in tumors banked at baseline.

VII. Evaluate EBV and HHV-8 gene expression patterns in positive tumors banked at baseline.

OUTLINE: This is a phase I, dose-escalation study of vorinostat followed by a phase II study.

PHASE I: Patients receive vorinostat orally (PO) once daily (QD) on days 1-5; rituximab intravenously (IV) on day 1; etoposide IV over 24 hours, doxorubicin hydrochloride IV over 24 hours, and vincristine sulfate IV over 24 hours on days 1-4; prednisone PO daily on days 1-5; and cyclophosphamide IV over 1 hour on day 5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM A (VR-DA-EPOCH): Patients receive vorinostat, rituximab, etoposide, doxorubicin hydrochloride, vincristine sulfate, prednisone, and cyclophosphamide as in Phase I.

ARM B (DA-R-EPOCH): Patients receive rituximab, etoposide, doxorubicin hydrochloride, vincristine sulfate, prednisone, and cyclophosphamide as in Arm A.

In all arms, treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically documented diffuse large B-cell lymphoma (DLBCL) must meet at least 1 of the following risk criteria:

  * Age-adjusted International Prognostic Index (IPI) score: 2-3
  * Ki-67 >= 80%
  * Histologically, or cytologically documented activated B-cell-like (ABC, also known as post-GCB) subtype
  * Double hit variant, defined as having v-myc avian myelocytomatosis viral oncogene homolog (MYC) gene rearrangement in the presence of B-cell chronic lymphocytic leukemia (CLL)/lymphoma (BCL) 2 or BCL6 gene rearrangement

    * Other aggressive non-DLBCL non-Burkitt non-Hodgkin B-cell lymphoma variants as defined by the 2008 World Health Organization (WHO) classification, including rare CD20 negative B-cell lymphomas (i.e. plasmablastic lymphoma, and primary effusion lymphoma) are also eligible; grade 3B follicular lymphoma is also eligible as long as one the above risk criteria is met
* Participants who are untreated or who received a maximum of one (1) cycle of combination chemotherapy, including rituximab-containing regimens, prior are eligible; the start of previous chemotherapy cycle must occur at least 21 days prior to beginning treatment under this protocol, and such cycle will count towards the total maximum of 6 cycles under this study
* Documentation of HIV infection at any time prior to study entry; documentation may be molecular (detectable viral ribonucleic acid [RNA] by polymerase chain reaction [PCR]), serologic (positive enzyme-linked immunosorbent assay [ELISA] and positive Western blot), or other federally approved licensed HIV test; prior documentation of HIV seropositivity is acceptable
* All stages of disease
* Measurable or non-measurable tumor parameter(s); non-measurable tumor parameters are defined as not having bidimensional measurements (e.g., gastric or marrow involvement), but can be followed for response by other diagnostic tests such as gallium, positron emission tomography (PET) imaging, and/or bone marrow biopsy
* Performance status (PS) 0, 1, or 2 per the Eastern Cooperative Oncology Group (ECOG) performance status scale (Karnofsky performance score >= 50%)
* Able to provide informed consent
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN), unless elevated secondary to lymphomatous involvement of liver or biliary system, or due to other HIV medications (e.g., indinavir, tenofovir, or atazanavir); for direct bilirubin > 1.2 due to hepatic involvement by tumor for the initial dose of EPOCH drug adjustment
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times ULN (unless elevated due to secondary lymphomatous involvement of the liver)
* Negative for hepatitis B, or if infected with hepatitis B, receiving anti-hepatitis B therapy; all participants will be required to be screened for hepatitis B and C; per Infectious Disease Society of America (IDSA) and American Association for the Study of Liver Diseases (AASD) guidelines, those participants that show no immunity, defined by the lack of hepatitis B surface antibody, and show evidence of chronic infection (i.e. hepatitis B surface antigen positive [HBsAg+], hepatitis B core antibody positive [HBcore+], hepatitis surface antibody negative [HBsAB-]) will be required to be on anti-hepatitis B therapy, during the study, in order to be eligible; participants will be permitted to enroll in the study provided liver function tests meet criteria, and there is no evidence of cirrhosis; the exact hepatitis B therapy will be at the discretion of the infection disease specialist or investigator; however all participants who present with acute hepatitis B or show normal transaminases and are HBsAg+ and immunoglobulin (Ig)M+ for hepatitis core antigen will not be eligible for trial enrollment; participants who are hepatitis C antibody positive, with or without a positive hepatitis C RNA level, will be permitted to enroll in the study provided liver function tests meet criteria, and have no evidence of cirrhosis; participants diagnosed with hepatitis C less than 6 months from trial enrollment, will be considered to have acute hepatitis C and will be excluded from study unless hepatitis (hep) C viral load is undetectable
* Creatinine clearance >= 60 mL/min, unless secondary to renal involvement by lymphoma; for creatinine clearance < 50 mL/min due to kidney involvement by tumor
* Granulocytes/absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelets >= 75,000/mm^3 (unless these parameters are abnormal secondary to lymphomatous involvement of bone marrow); all participants must cease colony-stimulating factor therapy at least 24 hours prior to institution of cycle 1 chemotherapy
* Left ventricular ejection fraction (LVEF) that is at or above the lower institutional limits of normal, as assessed by multiple gated acquisition (MUGA) scan or echocardiogram within the 6 weeks prior to registration
* Concurrent radiation, with or without steroids, or steroids alone for emergency conditions secondary to lymphoma (i.e. cord compression, etc.) will be permitted
* Female participants must have a negative pregnancy test within 7 days of entering into the study; both men and women of child bearing potential must agree to use adequate methods of contraception for the duration of the treatment; women must avoid pregnancy, and men must avoid fathering children while in the study and for 6 months following the last study drug treatment
* Participants on an antiretroviral regimen should be receiving treatment that is in accordance with the current International acquired immune deficiency syndrome (AIDS) Society guidelines; the specific agents are at the discretion of the investigator and use of agents currently available on an expanded access basis is allowed but use of experimental antiretroviral agents or those containing zidovudine (including Combivir and Trizivir) are prohibited; changes to highly active anti-retroviral therapy (HAART) therapy may be made if medically necessary (toxicity, failure of regimen, etc.); antiretroviral naïve participants: participants who are not on HAART at study entry MUST begin therapy (utilizing the above guidelines) AFTER one cycle of chemotherapy has been completed under protocol; changes to HAART therapy may be made if medically necessary (toxicity, failure of regimen, etc.); concurrent therapy with zidovudine or a zidovudine-containing regimen (including Combivir and Trizivir) will be prohibited until 2 months following the participant's completion of chemotherapy as part of this protocol; the use of cobicistat (e.g., Tybost), or cobicistat containing single tablet regimens (e.g., Stribild) is prohibited during concurrent chemotherapy under this protocol; participants taking cobicistat or cobicistat-containing single table regimens must switch to a different agent or regimen prior to enrollment, and will remain on the regimen until at least 2 months following treatment discontinuation; Cobicistat is a pure and potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitor and has the potential to increase the area under the curve (AUC) of CYP3A4 substrates; therefore, both vincristine and doxorubicin would have the potential for drug drug interaction (DDI) with cobicistat since they are CYP3A4 substrates
* Participants already receiving erythropoietin or colony-stimulating factor therapy are eligible for participation, although the latter must be discontinued at least 24 hours prior to receiving chemotherapy
* Participants must be able to swallow oral medications

Exclusion Criteria:

* Participants who have received more than one (1) prior cycle of chemotherapy similar to cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone (CHOP) or EPOCH with or without rituximab
* Absolute CD4 count of < 50 cells/ mm^3
* Presence of second active tumor, other than non-melanoma skin cancer, carcinoma in situ of the cervix, or Kaposi's sarcoma (KS) that requires systemic therapy
* Central nervous system (CNS) involvement by lymphoma including parenchymal brain or spinal cord lymphoma or known presence of leptomeningeal disease prior to registration
* Participants with viral hepatitis who do not meet the criteria will not be eligible; all participants who present with acute hepatitis B including those with normal transaminases who are HBsAg+ and IgM + for hepatitis core antigen will not be eligible; participants who are hepatitis B core antibody positive are eligible only if they start or are on prophylactic therapy; a hepatitis B viral load should be confirmed negative on all participants who are hepatitis B core antibody positive, but hepatitis B antigen negative; participants refusing to take any anti-hepatitis B therapy during study will also be excluded; participants diagnosed with hepatitis C are eligible if they meet criteria
* Pregnant women or nursing mothers
* ECOG performance score >= 3 (Karnofsky performance status [KPS] < 50%)
* Expected survival < 2 months
* Unable to comply with the requirements of the protocol, or unable to provide adequate informed consent in the opinion of the principal investigator
* Serious, ongoing, non-malignant disease or infection, which in the opinion of the investigator and/or the sponsor would compromise other protocol objectives; participants with active opportunistic infections are ineligible
* Major surgery, other than diagnostic surgery, occurring 4 weeks prior to study entry; splenectomy will not be considered an exclusionary major surgery
* Rituximab therapy within the 12 months prior to study entry; participants treated with rituximab within 12 months prior to study registration are eligible only if it was given for indications other than the treatment of aggressive lymphoma
* Prior cytotoxic chemotherapy or radiotherapy for this lymphoma
* History of cutaneous or mucocutaneous reactions, or diseases in the past, due to any cause, severe enough to cause hospitalization or an inability to eat or drink for > 2 days; this exclusion relates to the long-term possibility of severe cutaneous or mucocutaneous reactions to rituximab that might occur at increased frequency in participants who have had severe skin disease or reactions in the past
* Use of zidovudine or cobicistat as part of the HAART regimen (a drug substitution at the time of study entry is allowed)
* Any acute, inter-current infection that may interfere with planned protocol treatment; participants with mycobacterium avium will not be excluded from study entry; chronic therapy with potentially myelosuppressive agents is allowed provided that entry hematologic criteria are met
* Myocardial infarction (MI) within 6 months prior to study entry, New York Heart Association (NYHA) class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
* Participants should not have taken valproic acid or another histone deacetylase inhibitor for at least 2 weeks prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-10-06 (Actual); Primary Completion 2016-11-12 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Ramos, Principal Investigator — AIDS Malignancy Consortium
Locations (35):
- United States (35):
  - Jackson Hospital and Clinic, Montgomery, Alabama
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Center for Clinical AIDS Research and Education, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - San Diego VA Medical Center, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Stroger Hospital of Cook County MBCCOP, Chicago, Illinois
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Washington University - Jewish, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Thomas Street Clinic, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Ramos JC, Sparano JA, Chadburn A, Reid EG, Ambinder RF, Siegel ER, Moore PC, Rubinstein PG, Durand CM, Cesarman E, Aboulafia D, Baiocchi R, Ratner L, Kaplan L, Capoferri AA, Lee JY, Mitsuyasu R, Noy A. Impact of Myc in HIV-associated non-Hodgkin lymphomas treated with EPOCH and outcomes with vorinostat (AMC-075 trial). Blood. 2020 Sep 10;136(11):1284-1297. doi: 10.1182/blood.2019003959. PMID 32430507

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: VR-DA-EPOCH, Dose Level 1: Arm A (VR-DA-EPOCH) with Vorinostat at 300 mg once a day on days 1-5 of a cycle (Phase I Dose Level 1)
- Phase I: VR-DA-EPOCH, Dose Level 2: Arm A (VR-DA-EPOCH) with Vorinostat at 400 mg once a day on days 1-5 of a cycle (Phase I Dose Level 2)
- Phase I: VR-CHOP, Dose Level 1: Arm C (VR-CHOP) with Vorinostat at 300 mg once a day on days 1-5 of a cycle (Phase I Dose Level 1 for low risk participants). This arm was discontinued due to low accrual.
- Phase II: VR-DA-EPOCH: Arm A (VR-DA-EPOCH) at the recommended phase II dose of Vorinostat (300 mg once a day for days 1-5 of a cycle)
- Phase II: DA-R-EPOCH: Arm B (DA-R-EPOCH), which is the same treatment as Arm A, but without Vorinostat
Period: Phase I: VR-DA-EPOCH, Dose Level (DL) 1
Arm/Group | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: VR-CHOP, Dose Level 1 | Phase II: VR-DA-EPOCH | Phase II: DA-R-EPOCH
Started | 3 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase I: VR-DA-EPOCH, DL 2
Arm/Group | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: VR-CHOP, Dose Level 1 | Phase II: VR-DA-EPOCH | Phase II: DA-R-EPOCH
Started | 0 | 7 | 0 | 0 | 0
Completed | 0 | 6 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Ineligible | 0 | 1 | 0 | 0 | 0
Period: Phase I: VR-DA-EPOCH, DL 1 (De-escalate)
Arm/Group | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: VR-CHOP, Dose Level 1 | Phase II: VR-DA-EPOCH | Phase II: DA-R-EPOCH
Started | 4 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Ineligible | 1 | 0 | 0 | 0 | 0
Period: Phase I: VR-CHOP, DL 1
Arm/Group | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: VR-CHOP, Dose Level 1 | Phase II: VR-DA-EPOCH | Phase II: DA-R-EPOCH
Started | 0 | 0 | 2 | 0 | 0
Completed | 0 | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Noncompliant (Cycle 1 not complete) | 0 | 0 | 1 | 0 | 0
Period: Phase II: Randomized Groups
Arm/Group | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: VR-CHOP, Dose Level 1 | Phase II: VR-DA-EPOCH | Phase II: DA-R-EPOCH
Started | 0 | 0 | 0 | 45 | 46
Completed | 0 | 0 | 0 | 33 | 36
Not Completed | 0 | 0 | 0 | 12 | 10
Not completed — Death | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 2
Not completed — Ineligible | 0 | 0 | 0 | 0 | 1
Not completed — Disease progression/relapse on treatment | 0 | 0 | 0 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Eligible participants completing at least one cycle of treatment; 3 ineligible participants and 1 participant not completing one cycle of Phase I treatment were not included.
Groups:
- Phase II, V+DA-EPOCH: Arm A (VR-DA-EPOCH) at the recommended phase II dose of Vorinostat (300 mg once a day for days 1-5 of a cycle)
- Phase II, DA-R-EPOCH: Arm B (DA-R-EPOCH), which is the same treatment as Arm A, but without Vorinostat
- Total: Total of all reporting groups
Arm/Group | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: VR-CHOP, Dose Level 1 | Phase II, V+DA-EPOCH | Phase II, DA-R-EPOCH | Total
Number analyzed (Participants) | 6 | 6 | 1 | 45 | 45 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (12.4) | 50.4 (10.1) | 59.5 (0) | 49.2 (10.1) | 45 (9.2) | 47.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 6 | 0 | 7
  Male | 6 | 5 | 1 | 39 | 45 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 14 | 13 | 29
  Not Hispanic or Latino | 5 | 5 | 1 | 29 | 30 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 12 | 8 | 22
  White | 4 | 6 | 1 | 23 | 31 | 65
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 8 | 4 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 1 | 45 | 45 | 103

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) as Assessed by Response Evaluation Criteria in Solid Tumors (Phase II)
Description: Percentage of participants with complete response as assessed by Response Evaluation Criteria in Solid Tumors (Phase II) according to treatment arm. Participants are planned to be treated for a total of 6 cycles (21 day cycle length). Participants with CR after Cycle 4 will receive two additional cycles of chemotherapy and complete 6 cycles of chemotherapy. Participants who achieve a partial response (PR) only after Cycle 4 may continue on protocol therapy or they may be removed from the study at the AMC discretion of the physician (local Principal Investigator). Participants with stable disease after 4 cycles (i.e., who did not achieve at least a PR) or progressive disease at any time will be removed from study.
  In phase II, there are two arms: Vorinostat RPTD+rituximab-DA-EPOCH arm (VR-DA-EPOCH) and Rituximab-DA-EPOCH arm (DA-R-EPOCH).
Time Frame: Up to 6 months
Population: Reviewed responses from participants who completed at least one cycle of treatment. In phase II, there are two arms: Vorinostat RPTD+rituximab-DA-EPOCH arm (VR-DA-EPOCH) and Rituximab-DA-EPOCH arm (DA-R-EPOCH).
  In phase I, patients in DA-R-EPOCH were not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: VR-DA-EPOCH | Phase II: DA-R-EPOCH
Number analyzed (Participants) | 40 | 42
percentage of participants | 67.5 [50.9 to 81.4] | 76.2 [60.6 to 88.0]

2. Primary Outcome: Percentage of Participant Experiencing Adverse Events (AEs) for Each Treatment Arm as Assessed by Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0) (Phase II)
Description: The percentage of participants with AEs and their worst severity will be tabulated for each treatment arm. If a participant has more than one AE, the most severe AE is analyzed. All adverse events will be assessed by the investigator from the first dose of protocol therapy through the post-treatment discontinuation visit. Participants are planned to be treated for a total of 6 cycles (21 day cycle length), or roughly 4 months. After this evaluation, assessment and reporting of AEs will only be required for all grade 5 AEs and any serious AE (SAE) that the investigator considers related to protocol therapy.
Time Frame: Up to 5 years
Population: Eligible randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Phase II: VR-DA-EPOCH | Phase II: DA-R-EPOCH
Number analyzed (Participants) | 45 | 45
percentage of participants
  Death | 28.9 | 20.0
  Life-threatening | 37.8 | 28.9
  Severe | 20.0 | 31.1
  Moderate | 8.9 | 17.8
  Mild | 2.2 | 0

3. Primary Outcome: Recommended Phase II Dose of Vorinostat Determined According to Dose-limiting Toxicities Graded Using Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0) (Phase I)
Description: Recommended phase II dose of vorinostat is defined as the dose level at which 0/6 or 1/6 subjects experience dose limiting toxicity (DLT) with the next higher dose having at least 2/3 or 2/6 subjects encountering DLT (Phase I). Toxicities will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. Using a 3+3 design, the recommended phase II dose is defined as the level at which 0/6 or 1/6 patients experiences at dose-limiting toxicity in the first cycle.
Time Frame: 21 days
Population: Eligible Phase I Arm A (VR-DA-EPOCH) participants who completed at least 1 cycle of treatment. This arm includes participants treated at 300 mg once a day (n=6) or 400 mg once a day (n=6) of Vorinostat for days 1-5.
Measure: Number; unit: Mg per day of Vorinostat
Groups:
- Phase I: VR-DA-EPOCH: Phase I, Arm A (VR-DA-EPOCH)
Arm/Group | Phase I: VR-DA-EPOCH
Number analyzed (Participants) | 12
Mg per day of Vorinostat | 300

4. Secondary Outcome: Change in CD8 Cell Counts (Phase I)
Description: Differences from baseline (specified follow-up assessment minus baseline) in absolute CD8 counts.
Time Frame: Baseline up to 12 months
Population: Eligible participants who returned for follow-up with evaluable data.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Groups:
- Phase I: VR-DA-EPOCH, Dose Level 1: Phase I, Arm A (VR-DA-EPOCH) with Vorinostat at 300 mg once a day on days 1-5 of a cycle (Phase I Dose Level 1)
- Phase I: VR-DA-EPOCH, Dose Level 2: Phase I, Arm A (VR-DA-EPOCH) with Vorinostat at 400 mg once a day on days 1-5 of a cycle (Phase I Dose Level 2)
Arm/Group | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: VR-CHOP, Dose Level 1
Number analyzed (Participants) | 4 | 5 | 1
cells/mm^3
  End of cycle 2 | 35.5 [-348.5 to 356.5] | -115 [-162 to 75] | -172 [-172 to -172]
  Treatment discontinuation | -164.5 [-962.5 to 198.5] | 211 [18 to 359] | -81 [-81 to -81]
  6-month follow-up: number analyzed (Participants) | 3 | 5 | 1
  6-month follow-up | -56 [-177 to 443] | 275 [-152 to 728] | -16 [-16 to -16]
  12-month follow-up: number analyzed (Participants) | 1 | 5 | 1
  12-month follow-up | 604 [604 to 604] | 154 [-97 to 692] | 128 [128 to 128]

5. Secondary Outcome: Changes in Absolute CD4 Cell Counts (Phase I)
Description: Differences from baseline (specified follow-up assessment minus baseline) in absolute CD4 counts.
Time Frame: Baseline up to 12 months
Population: Eligible participants who completed at least 1 cycle of treatment with evaluable data.
Measure: Median (Inter-Quartile Range); unit: cell/mm^3
Groups:
- Phase I: VR-CHOP, Dose Level 1: Phase I, Arm C (VR-CHOP) with Vorinostat at 300 mg once a day on days 1-5 of a cycle (Phase I Dose Level 1 for low risk participants). This arm was discontinued due to low accrual.
Arm/Group | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: VR-CHOP, Dose Level 1
Number analyzed (Participants) | 6 | 6 | 1
cell/mm^3
  End of cycle 2 | 92 [9 to 143] | -9 [-41 to 49] | -218 [-218 to -218]
  Treatment discontinuation: number analyzed (Participants) | 6 | 5 | 1
  Treatment discontinuation | -39 [-53 to 56] | -29 [-32 to 41] | -190 [-190 to -190]
  6-month follow-up: number analyzed (Participants) | 3 | 5 | 1
  6-month follow-up | 76 [75 to 181] | 31 [-9 to 45] | -175 [-175 to -175]
  12-month follow-up: number analyzed (Participants) | 1 | 5 | 1
  12-month follow-up | 169 [169 to 169] | 31 [-16 to 104] | -84 [-84 to -84]

6. Secondary Outcome: Changes in Epstein-Barr Virus (EBV) Viral Load
Description: Differences from baseline (specified follow-up assessment minus baseline) in EBV viral load.
Time Frame: Baseline up to 12 months
Population: Median Change from the baseline and IQR were calculated. The measurement unit is IU/mL.
Measure: Median (Inter-Quartile Range); unit: IU/mL
Groups:
- Phase II, VR-DA-EPOCH: Arm A (VR-DA-EPOCH) at the recommended phase II dose of Vorinostat (300 mg once a day for days 1-5 of a cycle).
- Phase I: VR-DA-EPOCH, Dose Level 1: Arm A (VR-DA-EPOCH) with Vorinostat at 300mg once a day on days 1-5 of a cycle (Phase I dose Level 1)
- Phase I: VR-DA-EPOCH, Dose Level 2: Arm A (VR-DA-EPOCH) with Vorinostat at 400mg once a day on days 1-5 of a cycle (Phase I dose Level 1)
Arm/Group | Phase II, VR-DA-EPOCH | Phase II, DA-R-EPOCH | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: VR-CHOP, Dose Level 1
Number analyzed (Participants) | 16 | 19 | 1 | 1 | 0
IU/mL
  End of Cycle 2 | -0.61 [-104.1 to 0] | 0 [-0.61 to 0] | 0 [0 to 0] | -2436.1 [-2436.1 to -2436.1] |
  At treatment discontinuation: number analyzed (Participants) | 11 | 18 | 1 | 1 | 0
  At treatment discontinuation | -2.9 [-449.6 to -0.14] | -0.28 [-1.9 to 0] | 0 [0 to 0] | -1.92 [-1.92 to -1.92] |
  6-month follow-up: number analyzed (Participants) | 6 | 10 | 1 | 1 | 0
  6-month follow-up | -1.55 [-2.98 to 0] | 0 [-4.87 to 4.07] | 0 [0 to 0] | -1.92 [-1.92 to -1.92] |
  12-month follow-up: number analyzed (Participants) | 8 | 11 | 1 | 1 | 0
  12-month follow-up | -0.56 [-228.2 to -0.07] | -2.7 [-4.75 to 0] | 0 [0 to 0] | -1.15 [-1.15 to -1.15] |

7. Secondary Outcome: Changes in Human Herpes Virus (HHV)-8 Viral Load
Description: Differences from baseline (specified follow-up assessment minus baseline) in (HHV)-8 viral load.
Time Frame: Baseline up to 12 months
Population: Outcome measure is the difference between the baseline and specific time points (End of Cycle 2, Treatment discontinuation, 6-month, and 12-month follow-ups.
  Only a few differences can be calculated.
Measure: Median (Inter-Quartile Range); unit: copies per 100uL
Arm/Group | Phase II: VR-DA-EPOCH | Phase II: DA-R-EPOCH
Number analyzed (Participants) | 1 | 2
copies per 100uL
  End of Cycle 2: number analyzed (Participants) | 0 | 0
  At treatment discontinuation: number analyzed (Participants) | 0 | 1
  At treatment discontinuation |  | 0 [0 to 0]
  6-month follow-up: number analyzed (Participants) | 0 | 1
  6-month follow-up |  | 0 [0 to 0]
  12-month follow-up: number analyzed (Participants) | 1 | 1
  12-month follow-up | 0 [0 to 0] | 0 [0 to 0]

8. Secondary Outcome: Changes in Human Immunodeficiency Virus (HIV) Viral Load
Description: Differences from baseline (specified follow-up assessment minus baseline) in HIV viral load. Undetectable viral load results were treated as 0 values.
Time Frame: Baseline up to 12 months
Population: Phase II participants who returned for follow-up with evaluable data.
Measure: Median (Inter-Quartile Range); unit: median change in copies per mL
Arm/Group | Phase II: VR-DA-EPOCH | Phase II: DA-R-EPOCH
Number analyzed (Participants) | 42 | 41
median change in copies per mL
  End of Cycle 2 | -20 [-22607 to 0] | -25 [-3308 to 0]
  At treatment discontinuation: number analyzed (Participants) | 42 | 40
  At treatment discontinuation | -87 [-28176 to 0] | -22.5 [-1962 to 4.5]
  6-month follow-up: number analyzed (Participants) | 42 | 26
  6-month follow-up | -20 [-24703 to 0] | -18 [-3258 to 0]
  12-month follow-up: number analyzed (Participants) | 42 | 23
  12-month follow-up | 0 [-22656 to 20] | -20 [-3361 to 0]

9. Secondary Outcome: Event-free Survival (EFS) (Phase II)
Description: The percentage of participants surviving without events (relapse or death) one year after starting treatment.
Time Frame: 1 year
Population: Eligible randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: VR-DA-EPOCH | Phase II: DA-R-EPOCH
Number analyzed (Participants) | 45 | 45
percentage of participants | 75.6 [63.0 to 88.1] | 82.2 [71.1 to 93.4]

10. Secondary Outcome: Overall Survival (OS) (Phase II)
Description: The percentage of participants surviving one year after starting treatment.
Time Frame: 1 year
Population: Eligible randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: VR-DA-EPOCH | Phase II: DA-R-EPOCH
Number analyzed (Participants) | 45 | 45
percentage of participants | 77.6 [65.3 to 89.8] | 86.7 [76.7 to 96.6]

11. Secondary Outcome: Change in Plasma Associated Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) (Phase I)
Description: as for outcome 8
Time Frame: Baseline up to 12 months
Population: Eligible participants who returned for follow-up with evaluable data.
Measure: Median (Inter-Quartile Range); unit: copies per milliliter
Arm/Group | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: VR-CHOP, Dose Level 1
Number analyzed (Participants) | 6 | 6 | 1
copies per milliliter
  End of cycle 2 | -14518 [-54352 to 0] | -12.5 [-66 to 0] | 28 [28 to 28]
  Treatment discontinuation: number analyzed (Participants) | 6 | 5 | 1
  Treatment discontinuation | -4517 [-55116 to 0] | 0 [-88 to 49] | 0 [0 to 0]
  6-month follow-up: number analyzed (Participants) | 3 | 5 | 1
  6-month follow-up | -55116 [-282977 to 0] | 0 [-88 to 0] | 0 [0 to 0]
  12-month follow-up: number analyzed (Participants) | 1 | 5 | 1
  12-month follow-up | 0 [0 to 0] | 0 [-88 to 0] | 0 [0 to 0]

12. Secondary Outcome: Pharmacokinetic Clearance (Phase I)
Description: Serial plasma samples for pharmacokinetic analysis were collected at 24-48, 48-72, and 72-96 hours after the start of the first chemotherapy infusion. Doxorubicin, etoposide, and vincristine concentrations were determined using a validated liquid chromatography-tandem mass spectrometry method. The clearance was determined by dividing the drug-infusion rate by the steady-state concentrations, which was the average of the three time points.
Time Frame: 24-48, 48-72, and 72-96 hours after the start of the first chemotherapy infusion
Population: Phase I participants with evaluable pharmacokinetic data
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: VR-CHOP, Dose Level 1
Number analyzed (Participants) | 6 | 5 | 0
Liter/hour
  Doxorubicin | 78.6 (48.0) | 76.0 (47.9) |
  Etoposide | 3.0 (1.6) | 2.4 (0.7) |
  Vincristine | 22.4 (10.2) | 16.8 (8.9) |

13. Secondary Outcome: Tumor Response (Phase I)
Description: The percentage of participants whose best tumor response is complete response (CR) or partial response (PR). Based on clinical, radiologic (CT), and pathologic criteria, CR requires 1) complete disappearance of all detectable disease and disease-related symptoms if present before therapy, 2) bone marrow aspirate and biopsy to confirm a CR if initially positive or if clinically indicated by new abnormalities in the peripheral blood counts or blood smear, 3) negative PET results, depending on typically, variably, or unknown pre-treatment FDG status, and 4) spleen and/or liver, if considered to be enlarged before therapy on physical examination or CT scan, not being palpable on physical examination and considered normal size by imaging studies, and nodules related to lymphoma disappeared. PR includes 1) ≥50% decrease in sum of product of diameters (SPD), 2) no increase in size of nodes, liver, or spleen, 3) splenic/hepatic nodules regressed by ≥ 50% SPD, 4) no new sites of disease
Time Frame: Up to 2 years post treatment
Population: Eligible participants who completed at least 1 cycle of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase I: Arm C (VR-CHOP) Dose Level 1: Arm C (VR-CHOP) with Vorinostat at 300 mg once a day on days 1-5 of a cycle (Phase I Dose Level 1 for low risk participants). This arm was discontinued due to low accrual.
Arm/Group | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: Arm C (VR-CHOP) Dose Level 1
Number analyzed (Participants) | 6 | 6 | 1
percentage of participants
  Complete response | 83.3 [35.9 to 99.6] | 83.3 [35.9 to 99.6] | 100 [2.5 to 100]
  Partial Response | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 0 [0 to 97.5]

ADVERSE EVENTS:
Time Frame: Up to 5 years. Participants are planned to be treated for a total of 6 cycles (21 day cycle length), or roughly 4 months. All adverse events will be assessed by the investigator from the first dose of protocol therapy through the post-treatment discontinuation visit. After this evaluation, assessment and reporting of AEs will only be required for all grade 5 AEs and any SAE that the investigator considers related to protocol therapy.
Groups:
- Phase II: DA-R-EPOCH: Arm B (DA-R-EPOCH), which is the same treatment as Arm A but without Vorinostat
Arm/Group | Phase I: VR-DA-EPOCH, Dose Level 1 | Phase I: VR-DA-EPOCH, Dose Level 2 | Phase I: VR-CHOP, Dose Level 1 | Phase II: VR-DA-EPOCH | Phase II: DA-R-EPOCH
All-Cause Mortality (participants affected / at risk) | 2/7 | 1/7 | 0/2 | 13/45 | 9/46
Serious Adverse Events (participants affected / at risk) | 5/7 | 3/7 | 0/2 | 25/45 | 21/46
Other Adverse Events (participants affected / at risk) | 7/7 | 6/7 | 2/2 | 43/45 | 43/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: VR-DA-EPOCH, Dose Level 1 (N=7) | Phase I: VR-DA-EPOCH, Dose Level 2 (N=7) | Phase I: VR-CHOP, Dose Level 1 (N=2) | Phase II: VR-DA-EPOCH (N=45) | Phase II: DA-R-EPOCH (N=46)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 10 | 8
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 2
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 0 | 3 | 2
Cardiac Disorders - Other, Specify (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 1
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Esophageal Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastric Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Intra-Abdominal Hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mucositis Oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Rectal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 3
Death Nos (General disorders) | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Multi-Organ Failure (General disorders) | 0 | 0 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Enterocolitis Infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infections And Infestations - Other, Specify (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Kidney Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Sepsis (Infections and infestations) | 1 | 0 | 0 | 3 | 3
Soft Tissue Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tooth Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 2 | 0
Neutrophil Count Decreased (Investigations) | 5 | 2 | 0 | 12 | 2
Platelet Count Decreased (Investigations) | 0 | 3 | 0 | 11 | 0
White Blood Cell Decreased (Investigations) | 5 | 0 | 0 | 5 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 7 | 4
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Nervous System Disorders - Other, Specify (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal And Urinary Disorders - Other, Specify (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal Colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Surgical And Medical Procedures - Other, Specify (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Thromboembolic Event (Vascular disorders) | 1 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: VR-DA-EPOCH, Dose Level 1 (N=7) | Phase I: VR-DA-EPOCH, Dose Level 2 (N=7) | Phase I: VR-CHOP, Dose Level 1 (N=2) | Phase II: VR-DA-EPOCH (N=45) | Phase II: DA-R-EPOCH (N=46)
Anemia (Blood and lymphatic system disorders) | 2 | 4 | 1 | 27 | 23
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 4 | 2
Watering Eyes (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 8 | 4
Anal Mucositis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 3 | 2 | 0 | 20 | 18
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 0 | 17 | 10
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 3
Gastrointestinal Disorders - Other, Specify (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3
Mucositis Oral (Gastrointestinal disorders) | 2 | 2 | 0 | 9 | 9
Nausea (Gastrointestinal disorders) | 6 | 3 | 1 | 20 | 22
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 10 | 9
Chills (General disorders) | 1 | 0 | 0 | 5 | 0
Edema Limbs (General disorders) | 0 | 0 | 0 | 10 | 4
Fatigue (General disorders) | 2 | 2 | 2 | 18 | 13
Fever (General disorders) | 0 | 2 | 0 | 8 | 2
Flu Like Symptoms (General disorders) | 0 | 1 | 0 | 0 | 0
General Disorders And Administration Site Conditions - Other, Specify (General disorders) | 0 | 0 | 0 | 2 | 3
Infusion Related Reaction (General disorders) | 1 | 0 | 0 | 1 | 2
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 2 | 3
Abdominal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Esophageal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infections And Infestations - Other, Specify (Infections and infestations) | 0 | 0 | 0 | 5 | 0
Mucosal Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 4
Nail Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Rhinitis Infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper Respiratory Infection (Infections and infestations) | 0 | 1 | 0 | 2 | 2
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 18 | 9
Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0 | 11 | 9
Aspartate Aminotransferase Increased (Investigations) | 1 | 1 | 0 | 15 | 10
Blood Bilirubin Increased (Investigations) | 1 | 0 | 0 | 4 | 2
Creatinine Increased (Investigations) | 0 | 0 | 0 | 4 | 4
Ggt Increased (Investigations) | 0 | 0 | 0 | 2 | 3
Lymphocyte Count Decreased (Investigations) | 1 | 3 | 1 | 20 | 19
Lymphocyte Count Increased (Investigations) | 0 | 1 | 0 | 0 | 2
Neutrophil Count Decreased (Investigations) | 4 | 2 | 0 | 24 | 19
Platelet Count Decreased (Investigations) | 4 | 3 | 1 | 27 | 19
Weight Loss (Investigations) | 1 | 1 | 0 | 3 | 0
White Blood Cell Decreased (Investigations) | 3 | 2 | 0 | 25 | 21
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 23 | 16
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 4
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 14 | 15
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 11 | 16
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 5
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 23 | 15
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 6 | 7
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 14 | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 7 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 4 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 4
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 3 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3
Cognitive Disturbance (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 6 | 5
Dysesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 9 | 17
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 3 | 3
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 4 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 1 | 0 | 12 | 20
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 5 | 3
Depression (Psychiatric disorders) | 0 | 0 | 0 | 4 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 5 | 7
Urinary Frequency (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 4
Urinary Tract Pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 3
Oligospermia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 4 | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 4 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 4 | 6
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 1
Hyperhidrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 2
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 4 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 4
Lymphedema (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 5 | 1

LIMITATIONS AND CAVEATS:
Experimental Arm C (VR-CHOP) was discontinued early in phase I due to low accrual; only 2 participants received VR-CHOP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less